CLINICAL TRIAL: NCT05453526
Title: Burden of Valvular Heart Diseases in an Ethnical/Racial Diverse Background of the United States: the Bronx-Valve Registry
Brief Title: The Bronx-Valve Registry
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13933
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Valvular Heart Disease
Keywords: valvular heart disease; race; ethnicity; diversity; mitral valve; aortic valve; tricuspid valve; pulmonary valve; stenosis; regurgitation; echocardiography
MeSH Terms: conditions — Heart Valve Diseases; Constriction, Pathologic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Race - American Indian or Alaska Native: Being identified as American Indian or Alaska Native
- Race - Asian: Being identified as Asian
- Race - Black or African-American: Being identified as Black or African-American
- Race - Native Hawaiian or Other Pacific Islander: Being identified as Native Hawaiian or Other Pacific Islander
- Race - White: Being identified as White
- Ethnicity - Spanish/Hispanic/Latino: Being identified as Spanish/Hispanic/Latino

SUMMARY:
The Bronx-Valve Registry is designed to collect and assess data on all patients with valvular diseases referred to Montefiore Medical Center for echocardiographic exams. Valvular heart disease (VHD) is a major focus of cardiovascular medicine, but limited data are available for racial and ethnic minorities. The aim was to assess the burden and clinical correlates of VHD in a highly diverse area of the United States.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in the general US population. Although the burden of valvular heart disease is increasing due to a rapidly aging population, patients can benefit from improved and more accessible imaging modalities, and novel minimally invasive treatments. However, medical knowledge and technological developments might not be generalizable to all patient backgrounds due to lack of diversity in scientific literature.

Historically, clinical trials testing new treatment modalities have lacked equitable inclusion of people coming from racial/ethnic minority groups. Similarly, epidemiological studies have focused on specific patient subsets with no direct comparisons with the other backgrounds. The Bronx county (New York, USA) is considered by the US Census as the most diverse area in the country, having the highest overwhelming concentration of non-white populations and being the only borough in all of New York City to be almost exclusively populated by non-white enclaves. These demographic characteristics make this county ideal to assess how the prevalence and the clinical correlates of valvular heart diseases might vary among diverse populations.

On this background, the objective of this registry is to assess the burden of valvular heart diseases and explore their clinical correlates in the most diverse area of the United States.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Undergoing transthoracic or transesophageal echocardiographic assessment at Montefiore Medical Center or affiliated institutions in the Bronx (NY, USA)

Exclusion Criteria:

* Age below 18 years old
* No available information regarding race or ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing echocardiographic assessment at Montefiore Medical Center (Bronx, NY, USA) will be included in this registry.
Sampling Method: Probability Sample
Enrollment: 330570 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Racial/ethnical based differences in baseline characteristics and valvular heart disease | Baseline
  Baseline characteristics among pre-defined racial/ethnical groups will be compared for each valvular heart disease
Prevalence of Valvular Heart Disease | Up to 10 years
  Prevalence of each valvular heart disease will be compared among pre-defined racial/ethnical groups
All-cause mortality | Up to 10 years
  All-cause mortality according to valvular heart disease and racial/ethnical group

CONTACTS AND LOCATIONS:
Overall Officials: Azeem Latib, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Echarte-Morales J, Scotti A, Bonnet G, Torrado J, Sturla M, Coisne A, Ludwig S, Barzallo D, Escabia C, Chandra A, Kodesh A, Aftab A, Granada JF, Ho EC, Jorde UP, Rodriguez CJ, Slipczuk L, Garcia MJ, Latib A. Racial and ethnic disparities in patients with severe tricuspid regurgitation: The Bronx-Valve registry. Int J Cardiol. 2025 Feb 15;421:132889. doi: 10.1016/j.ijcard.2024.132889. Epub 2024 Dec 6. PMID 39647784
- [Result] Scotti A, Sturla M, Echarte-Morales J, Ho EC, Millin A, Coisne A, Ludwig S, Leone PP, Rosiene J, Granada JF, Goldberg Y, Pu M, Jorde UP, Slipczuk L, Rodriguez CJ, Garcia MJ, Latib A. Burden of Valvular Heart Diseases in a Racially and Ethnically Diverse Population: The Bronx-Valve Registry. J Am Heart Assoc. 2025 Jan 21;14(2):e035378. doi: 10.1161/JAHA.124.035378. Epub 2025 Jan 16. PMID 39817520